CLINICAL TRIAL: NCT00552214
Title: Evaluation of a TMA Assay for the Screening of HIV-1 RNA, HCV RNA and HBV DNA in Human Blood Donor Plasma Specimens
Brief Title: Evaluation of HIV-1, HCV and HBV Blood Screening Tests With Human Blood Donor Specimens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ULT-001-TW1-Amendment 1.1
Record Dates: First submitted 2007-10-30; First posted 2007-11-01 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Screening for the Presence of HIV-1, RNA and HBV DNA in Blood Donations
Keywords: Nucleic acid test; HIV-1; hepatitis; HBV; HCV; TMA; HIV Seronegativity
MeSH Terms: conditions — Hepatitis | interventions — Hematologic Tests

ARMS (1):
- Human Blood Donor Plasma Specimens (Other)
  Interventions: Device: Blood test

INTERVENTIONS:
Device: Blood test — Screening of HIV-1 RNA, HCV RNA and HBV DNA in Human Blood Donor Plasma Specimens

SUMMARY:
The purpose of this study is to validate the performance characteristics of an assay that tests for HIV-1, HCV and HBV on an automated blood bank instrument for registration submission.

ELIGIBILITY:
Inclusion Criteria:

* An acceptable blood donation health history and an EIA negative donation sample result with licensed EIA procedures in routine use at each facility

Exclusion Criteria:

* A positive (reactive) HIV and/or HCV and/or HBV test

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10290 (Actual)
Dates: Start 2007-08-08; Primary Completion 2008-07-01 (Actual); Study Completion 2008-07-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity | 01 August 2007 to 31 December 2007

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Grifols Biologicals, LLC
Locations (1):
- Taipei Blood Center Taiwan Blood Service Foundation (TBSF), Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Novartis results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2615